CLINICAL TRIAL: NCT01856582
Title: Post Transplant CD34+ Selected Stem Cell Infusion to Augment Graft Function in Children With Primary Immunodeficiency Diseases and Bone Marrow Failure Syndromes
Brief Title: CD34+ Stem Cell Infusion to Augment Graft Function
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CliniMACS CD34 Reagent System was FDA approved for clinical use; therefore, patients were treated clinically.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hoxworth Blood Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-2344
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2018-12

CONDITIONS: Waning Donor Chimerism; Waning Immune Function; Primary Immunodeficiency Disease(s); Bone Marrow Failure
Keywords: Primary Immunodeficiency Disease(s); Mixed Donor Chimerism; bone marrow failure syndromes; allogeneic hematopoietic stem cell transplant (HSCT); children
MeSH Terms: conditions — Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD34+ selected stem cell infusion (Experimental): An infusion of selected CD34+ stem cells will be given without any preparative regimen.
  Interventions: Biological: CD34+

INTERVENTIONS:
Biological: CD34+ — CD34+ cells are selected using the CliniMACS System; without preparative regimen

SUMMARY:
The purpose of this study is to determine if infusing additional special donor cells will help to improve graft or immune function in previously transplanted children with immune deficiencies and bone marrow failures.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the usefulness of infusing purified CD34+ cells of donor origin in order to augment graft function in response to declining chimerism after initially performing an allogeneic hematopoietic stem cell transplant (HSCT) for children with primary immunodeficiency diseases. This protocol will be utilized for patients with waning mixed donor chimerism that is inadequate for correction of clinical condition or disease for which stem cell transplant was performed, or for augmentation of immune function. An infusion of selected CD34+ stem cells will be given without any preparative regimen. As the children eligible for this protocol have reduced immune function and pre-existing donor chimerism, we hypothesize that stem cells will be able to engraft and the infusion will augment graft function. This therapy serves as an alternative to a second stem cell transplant that is known to be associated with significant morbidity and mortality. CD34+ stem cells will be collected from the donor used for initial stem cell transplant. Cells will be T-cell depleted (TCD) by performing a CD34 selection using the CliniMACS device (Miltenyi Biotec) in order to prevent development of new or exacerbation of existing graft versus host disease (GVHD), as avoidance of GVHD in nonmalignant diseases is desirable. There is sufficient data showing that mixed donor chimerism is adequate for reverting disease phenotype in certain primary immunodeficiencies. Observations from Europe and CCHMC show that donor chimerism might be boosted by CD34+ stem cell infusion alone without any specific preparative regimen. This therapy is likely to be associated with low toxicity due to the absence of a preparative regimen and lack of exposure to fresh donor cells capable of initiating GVHD, and offers potential significant benefit.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this protocol, patients must have the following:

1. Primary immunodeficiency (e.g. SCID, Wiskott-Aldrich and/or other more rare conditions and other bone marrow failure syndromes) with prior allogeneic stem cell transplant.
2. Waning donor chimerism or immune function that is inadequate to correct their disease or clinical condition, for which primary transplant was given, as determined by their attending physician.
3. Available primary donor.
4. Must not have other organ dysfunction deemed by the attending physician to preclude this procedure.
5. Age < 35 years at time of transplant
6. One of the following must be true:

   * Patients must have evidence of persistent or recurrent immunodeficiency or thrombocytopenia.

-OR-

• Primary immunodeficiency disease with known potential to progress to malignant condition if untreated.

-OR-

• Debilitating secondary disease known to be a consequence of inadequate immune response to known agent or pathogen, uncontrollable by other available medical therapies (e.g. third patient described on page 5).

Exclusion Criteria:

1. Absence of an available original donor
2. Failure to sign consent form, or inability to undergo informed consent process
3. Pregnant or lactating female
4. Uncontrolled GVHD

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2010-10; Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Marsh, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Chandra S, Bleesing JJ, Jordan MB, Grimley MS, Khandelwal P, Davies SM, Edwards S, Leemhuis T, Marsh RA. Post-Transplant CD34+ Selected Stem Cell "Boost" for Mixed Chimerism after Reduced-Intensity Conditioning Hematopoietic Stem Cell Transplantation in Children and Young Adults with Primary Immune Deficiencies. Biol Blood Marrow Transplant. 2018 Jul;24(7):1527-1529. doi: 10.1016/j.bbmt.2018.03.013. Epub 2018 Mar 16. PMID 29555312

RESULTS

PARTICIPANT FLOW:
Groups:
- CD34+ Selected Stem Cell Infusion: A single infusion of selected CD34+ stem cells will be given without any preparative regimen. Stem cells will be depleted of T-cells using a CliniMACS CD34+ cell selection device and infused into the patient with a maximum T-cell dose of 5 x 10^4/kg. The minimum number of CD34+ cells that will be infused is 1x10^6/kg.
Period: Overall Study
Arm/Group | CD34+ Selected Stem Cell Infusion
Started | 23
Completed | 22
Not Completed | 1
Not completed — Died prior to Boost infusion | 1

BASELINE CHARACTERISTICS:
Arm/Group | CD34+ Selected Stem Cell Infusion
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Showed Successful Augmentation of Graft Function
Description: Successful augmentation of graft function achieved if donor chimerism is doubled compared to the value immediately pre-infusion at 12 months.
Time Frame: 12 months
Population: Selected data from this study was combined with a clinical retrospective study for analysis and published.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Selected Stem Cell Infusion
Number analyzed (Participants) | 22
Participants | 3

ADVERSE EVENTS:
Time Frame: All AEs were collected for 30 days post stem cell infusion. Protocol-defined AEs related to study treatment were followed for three years.
Arm/Group | CD34+ Selected Stem Cell Infusion
All-Cause Mortality (participants affected / at risk) | 3/23
Serious Adverse Events (participants affected / at risk) | 8/23
Other Adverse Events (participants affected / at risk) | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD34+ Selected Stem Cell Infusion (N=23)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Chronic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (2)
Hypotension (Cardiac disorders) | 2 (4)
Fever (General disorders) | 1 (1)
Multiorgan Failure (General disorders) | 2 (3)
Infection (Infections and infestations) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD34+ Selected Stem Cell Infusion (N=23)
Hemolysis (Cardiac disorders) | 1 (1)
Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT01856582/Prot_SAP_000.pdf